CLINICAL TRIAL: NCT06620016
Title: Diagnostic Role of Circulating microRNAs in Small Testicular Masses Suitable for Testis Sparing Surgery and Post-chemotherapy Residual Masses Suitable for Retroperitoneal Lymph Node Dissection.
Brief Title: Circulating microRNAs in Small Testicular Masses and Retroperitoneal Post-chemotherapy Residual Masses.
Acronym: SEARCH-1
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: SEARCH-1
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-09

CONDITIONS: Testicular Cancer
MeSH Terms: conditions — Testicular Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: Small testicular mass suitable for testis sparing surgery.
  Interventions: Diagnostic Test: Circulating microRNAs.
- B: Retroperitoneal post-chemotherapy residual mass suitable for retroperitoneal lymph node dissection.
  Interventions: Diagnostic Test: Circulating microRNAs.

INTERVENTIONS:
Diagnostic Test: Circulating microRNAs. — Pre and post-surgery evaluation of peripheral blood circulating microRNAs levels.

SUMMARY:
The purpose of this study is to evaluate the diagnostic performance of circulating microRNAs in detecting the presence of germ cell cancer in patients with small testicular mass or retroperitoneal post-chemotherapy residual mass and suitable for testis sparing surgery and retroperitoneal lymph node dissection, respectively.

ELIGIBILITY:
COHORT A:

Inclusion Criteria:

* Age >= 18 years
* Single testicular lesion, with < 2 cm diameter and < 30 % testicular volume involvement;
* Negative Serum Tumour Markers;
* Suitable for testis sparing surgery;
* Informed consent.

Exclusion Criteria:

* None

COHORT B:

Inclusion Criteria:

* Age >= 18 years
* Single/multiple post-chemotherapy retroperitoneal lymph node lesion, with > 1 cm (non seminomatous) / > 3 cm (seminomatous) diameter in patients with previous testicular germ cell primary tumour;
* Negative Serum Tumour Markers;
* Suitable for retroperitoneal lymph node dissection;
* Informed consent.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All males >= 18 yo with small testicular mass suitable for testis sparing surgery or post-chemotherapy germ cell residual mass suitable for retroperitoneal lymph node dissection.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
MicroRNA's germ cell cancer detection (Cohort A) | Baseline.
  Preoperative circulating microRNA's diagnostic accuracy in detecting germ cell cancer in patients with small testicular mass and submitted to testis sparing surgery, using post-operative surgical specimen as reference.
MicroRNA's germ cell cancer detection (Cohort B) | Baseline.
  Preoperative circulating microRNA's diagnostic accuracy in detecting germ cell cancer in patients with post-chemotherapy residual mass and submitted to retroperitoneal lymph node dissection, using post-operative surgical specimen as reference.

SECONDARY OUTCOMES:
MicroRNA's germ cell cancer subtype detection (Cohort A + B) | Baseline.
  Preoperative circulating microRNA's diagnostic accuracy in detecting seminomatous and non-seminomatous germ cell cancer in patients with small testicular mass/post-chemotherapy residual mass and submitted to testis sparing surgery/retroperitoneal lymph node dissection, using post-operative surgical specimen as reference.
MicroRNA's vs Frozen Section Examination's germ cell cancer detection (Cohort A) | Baseline.
  Comparison between preoperative circulating microRNA and Frozen Section Examination in detecting germ cell cancer in patients with small testicular mass and submitted to testis sparing surgery, using post-operative surgical specimen as reference.
MicroRNA's disease recurrence/persistence detection (Cohort A + B) | Week 4.
  Postoperative circulating microRNA's diagnostic accuracy in detecting disease recurrence/persistence in patients with small testicular mass/post-chemotherapy residual mass and submitted to testis sparing surgery/retroperitoneal lymph node dissection, using post-operative radiological imaging as reference.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna Policlinico di S. Orsola, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes